CLINICAL TRIAL: NCT01324986
Title: A Study on the Effectiveness of Laparoscopic Fundoplication on Extraesophageal Manifestations of Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Public Hospital Zell am See (Other)
Other Study IDs: Zell 03
Record Dates: First submitted 2011-03-27; First posted 2011-03-29 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-03

CONDITIONS: Extraesophageal Symptoms; Gastroesophageal Reflux Disease (GERD)
Keywords: extraesophageal symptoms of gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux

ARMS (2):
- Nissen fundoplication (Active Comparator)
  Interventions: Procedure: Laparoscopic anti-reflux surgery
- Toupet fundoplication (Active Comparator)
  Interventions: Procedure: Laparoscopic anti-reflux surgery

INTERVENTIONS:
Procedure: Laparoscopic anti-reflux surgery

SUMMARY:
Available data regarding the effectiveness of laparoscopic antireflux surgery on extraesophageal symptoms of gastroesophageal reflux disease (GERD) are scarce and mostly controversial. The aim of the present study was to evaluate the clinical effect of partial and total fundoplication on extraesophageal symptoms in a selected cohort of patients with GERD.

ELIGIBILITY:
Inclusion Criteria:

* persistent or recurrent symptoms despite continuous medical treatment, at least one typical reflux symptom (heartburn/ regurgitation/dysphagia/epigastric pain) and/or at least one atypical reflux symptom (cough/ asthma/hoarseness/distortion of taste), pathologic esophageal acid exposure as documented by a reflux-related DeMeester score ≥14.7, and symptom correlation ≥50%, and/or reflux episodes >73.

Exclusion Criteria:

* previous esophageal or gastric surgery, poor physical status (American Society of Anesthesiologists (ASA) scores III and IV) and pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- General Public Hospital Zell am See, Zell am See, Salzburg, Austria